CLINICAL TRIAL: NCT04474561
Title: Exploring the Use of a Reduced Sulfur Diet to Improve Disease Severity in Ulcerative Colitis: An 8-week Randomized Controlled Trial
Brief Title: Reduced Sulfur Diet in Ulcerative Colitis Patients
Acronym: UCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Maitreyi Raman, Clinical Associate Professor, Director Clinician Investigator Program (CIP), Medical Director Alberta's Collaboration of Excellence for Nutrition in Digestive Diseases (Ascend) , Medical Director Nutrition Services, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REB16-2491
Record Dates: First submitted 2020-07-13; First posted 2020-07-17 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Ulcerative Colitis; Diet Habit
MeSH Terms: conditions — Colitis, Ulcerative; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced sulfur diet intervention (INT) (Other): The INT group will receive conventional management plus a reduced sulfur diet and diet counselling by an RD. Implementation of the diet will be delivered directly by the RD and will provide each patient with an individualized plan. A reduced sulfur diet includes reducing foods, additives and beverages high in sulfate/sulfur.
  The reduced sulfur diet eating plan, resources on reduced sulfur eating, and RD counselling session will be designed and reviewed by experts in nutrition, dietary design, education resources and dietary behaviour change
  Interventions: Other: Reduced sulfur diet
- Conventional management (CM) (No Intervention): The CM group will receive one session with RD on reduced sulfur diet at the end of 8 weeks.CM groups will receive conventional management .

INTERVENTIONS:
Other: Reduced sulfur diet — A reduced sulfur diet includes reducing foods, food additives (e.g., carrageenan) and beverages high in sulfate/sulfur, limiting sulfur containing supplements, and consuming omega-3 fatty acid supplements to potentially help control overgrowth of sulfur-reducing bacteria in the colon. Omega-3 fatty acid intake for cardiovascular disease prevention should be around 500 mg/d23. After dietary assessment if patients are not meeting their required daily intake of 500 mg/d of Omega-3, the RD will recommend increased fish consumption to 200 g per week or 1 g/d of an Omega-3 supplement. This will ensure the daily recommended intake of 500 mg/d is being met to reduce the chances of a deficiency; however, a therapeutic dose for UC will not be recommended (i.e., > 4 g/d18).
  Arms: Reduced sulfur diet intervention (INT)

SUMMARY:
A)Background:

Approximately 44% of patients with Inflammatory bowel disease have Ulcerative colitis(UC) which is a lifelong, chronic disease, starting in early adulthood, where the colon becomes inflamed and ulcerated due to a complex interaction between genetics, altered immune function, and environmental factors2such as dietary intake. While the etiology of UC is not clear, it is hypothesized the abnormal immune response and chronic inflammation may be caused by dysbiosis of the intestinal microbiota and decreased epithelial barrier function. Substantial evidence suggests that higher than normal levels of hydrogen sulfide (H2S) in the colon plays a role in the etiology of UC. The higher levels of H2S and sulfate-reducing bacteria (SRB) found in the feces of patients with UC is likely caused by the reduced conversion of H2S to thiosulfate by rhodanese (thiosulfate transferase enzyme)12, and increased colonization or activity of SRB. For example, SRB has been identified as the predominant bacterial group in patients with UC compared to the minority group in healthy individuals, and SRB growth is stimulated by the presence of sulfur-rich amino acids. Dietary intervention may help to repair the dysbiosis existing in the microbiome of the patient with UC, but research about food and recurrence of UC is conflicting. Dietary components such as sulfur and sulfates also appear to play a role in the recurrence of UC; although a recent review of the relationship between sulfur-containing foods and UC calls for more randomized controlled trials (RCTs) examining a reduced sulfur diet in UC. With the body of evidence described above, there is a compelling reason to consider that sulfur and sulfate-containing foods contribute to developing severe UC. Thus, understanding how dietary modulation of sulfur intake within the context of UC impacts disease status is the focus of this proposal.

DETAILED DESCRIPTION:
A)Overview and Specific Aims:

Higher than normal levels of hydrogen sulfide (H2S) in the colon plays an important role in the etiology of ulcerative colitis (UC). Increased H2S impairs the colonic cell's ability to oxidize butyrate and other short-chain fatty acids required for cell nutrition. Sulfur in the human body is largely provided by diet; high intakes of sulfur and sulfate-containing foods have been found to be associated with an increased risk of recurrence of UC. Hence, it is only rational to identify whether foods high in sulfur or sulfate increase the risk of poor outcomes in UC. To our knowledge, there have been no studies investigating the impact of a reduced sulfur diet compared to conventional management on disease severity in patients with UC. Our main objectives are to identify if a reduced sulfur diet added to conventional management results in 1. improved disease severity, 2. reduced exposure of the host to sulfur-containing compounds, and 3. alterations in the microbiome of the patients. To achieve these objectives, we will randomly allocate the patients to either the conventional management (CM) or reduced sulfur diet intervention group (INT) and obtain the Mayo score, concentrations of fecal hydrogen sulphide (H2S), methanethiol (MT), and dimethyl sulphide (DMS), and urinary dimethyl sulfone (DM202) and 3-indoxyl sulfate and fecal microbiome at baseline and after 8 weeks. The INT group will also receive diet counselling by a registered dietician (RD).

B)Hypothesis:

A reduced sulfur diet would result in improved disease severity compared to conventional management in UC patients.

C)Objectives:

Primary objective:

1. To pilot-test the feasibility of a reduced sulfur diet added to conventional management with oral and/or topical 5-ASA ± corticosteroid therapy to improve disease severity, measured by a clinically meaningful improvement in Total Mayo Score & partial Mayo Score from baseline to week 8 compared to conventional management alone.

Secondary objectives:

1. To pilot-test the feasibility of a reduced sulfur diet added to conventional management with oral and/or 5-ASA ± oral corticosteroids to lower exposure of the host to sulfur-containing compounds from baseline to week 8 measured by fecal hydrogen sulphide (H2S), methanethiol (MT), and dimethyl sulphide (DMS), and; urinary dimethyl sulfone (DM202), and 3-indoxyl sulfate concentration compared to conventional management alone.
2. To examine the effect of a reduced sulfur diet on the microbiome of patients with UC.
3. To identify patient experience with a reduced sulfur diet using health related quality of life (HRQoL), and patient experience with chronic disease care measures.
4. To examine the effect of a reduced sulfur diet on inflammatory cytokines in patients with UC.

D) Methods

Study Design :

This pilot randomized controlled trial will have an 8-week interventional design that will take place at the University of Calgary (UofC).

Patient Recruitment:

Dr. Raman, the principal investigator, will oversee recruitment of eligible patients. In addition, Dr. Panaccione, Director of the IBD unit at the University of Calgary, and co-investigator for this study who along with the eight physicians associated with the IBD group at the University of Calgary will identify eligible study patients through dedicated outpatient IBD clinics and refer to Dr. Raman and the study coordinator for recruitment. The Calgary IBD unit assesses approximately 600 patients per month with at least 20 of them meeting eligibility criteria for this research project. All patients with UC in the IBD clinic who meet inclusion criteria will be approached for participation by the study coordinator after approval from their gastroenterologist.

Randomization of the patients:

After the patient consents to participate s/he will be randomly allocated to either the conventional management (CM) or intervention group (INT). Randomization will be performed using a computerised random number generator and group assignment will be concealed from the study coordinator enrolling patients until the time of assignment using sealed envelopes.

Intervention:

The INT group will receive conventional management plus a reduced sulfur diet and diet counselling by an RD. Implementation of the diet will be delivered directly by the RD and will provide each patient with an individualized plan. A reduced sulfur diet includes reducing foods, food additives (e.g., carrageenan) and beverages high in sulfate/sulfur associated with increased severity of UC consuming drinking water low in sulfate (can be as high as 500 mg/L in Alberta so identifying drinking water source is necessary)21, limiting sulfur containing supplements (e.g., chondroitin sulfate), and consuming omega-3 fatty acid supplements to potentially help control overgrowth of sulfur-reducing bacteria in the colon14. Omega-3 fatty acid intake for cardiovascular disease prevention should be around 500 mg/d23. In a representative Canadian population, average intake was 291 mg/d and 85% of adults were not meeting daily requirements23. After dietary assessment if patients are not meeting their required daily intake of 500 mg/d of Omega-3, the RD will recommend increased fish consumption to 200 g per week or 1 g/d of an Omega-3 supplement. This will ensure the daily recommended intake of 500 mg/d is being met to reduce the chances of a deficiency; however, a therapeutic dose for UC will not be recommended (i.e., > 4 g/d18). The CM group will receive one session with RD on reduced sulfur diet at the end of 8 weeks.

The reduced sulfur diet eating plan, resources on reduced sulfur eating, and RD counselling session will be designed and reviewed by experts in nutrition, dietary design, education resources and dietary behaviour change. Both the INT and CM groups will receive conventional management with visits to the clinic at 4 weeks to ensure completion of their 24-hour food recalls and food frequency questionnaires, and to discuss disease course with their physician.

ELIGIBILITY:
Inclusion Criteria

* Age ≥18 years.
* Currently experiencing a mild or moderate UC flare managed with either ≥1.2 grams of oral 5-ASA, topical 5-ASA, combination oral and topical 5-ASA with or without oral corticosteroid therapy or UC in remission, define by partial Mayo score < 3, treated with any 5-ASA preparation, or biologic therapies
* Ability to provide informed consent and willingness to undergo 2 endoscopic assessments if flare.

Exclusion Criteria:

* Experiencing a severe UC flare.
* Have any other major medical comorbidities (diabetes, active malignancy within the past 5 years, active infections, severe respiratory or cardiac disease, or acute or chronic kidney disease).
* Have a history of previous bowel surgery.
* Smokers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-04-20 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Mayo Score: Change is being assessed | Baseline and week -8
  Mayo score is used for patients with active disease.Mayo Score is one of the most commonly used indices of UC severity. Score ranges from 0-12 with a score ≤ 2.5 indicating remission. Mayo Score includes ratings of stool frequency, rectal bleeding, mucosal appearance at endoscopy and physician rating of disease activity. Higher score means worse outcomes.
  For the patients in remission disease activity will be measured using the non-invasive partial Mayo Score calculated at baseline and week 8. Partial Mayo score excludes mucosal appearance at endoscopy but includes stool frequency, rectal bleeding, and physician rating of disease .

SECONDARY OUTCOMES:
Fecal sulfate: Change is being assessed | Baseline, week-8
  Stool kits will be provided.Patients will be asked to defecate into a plastic bag approximately 15 mL of feces and close the bag immediately, expel any air present and then put in a standard home freezer (-20°C).Fecal samples will be analysed for sulfur-containing compounds using gas chromatography.
Urinary sulfate: Change is being assessed | Baseline, Week -8
  24-HR urine jar plain will be provided.Patient will be asked to store the 24-Hr urine sample in home freezer as well. Both the specimens will be transported to the lab within 7 days of collection in a Styrofoam container on an ice pack.Urinary dimethyl sulfone (DM202) and 3-indoxyl sulfate will be analysed using quantitative NMR spectroscopy.
Stool microbiome: Change is being assessed | Baseline, Week-8
  While the patient population will be clinically homogenous the changes in bacterial composition may vary over short periods of time.Fecal DNA will be used as input for the Illumina Nextera® XT DNA Sample Preparation Kit to construct indexed paired-end DNA libraries as previously described. A final constructed paired-end indexed library set is run on a Bioanalyzer 2100 using Agilent High Sensitivity DNA Kit to acquire library average size distribution (Agilent Technologies, Santa Clara). Final libraries are quantified using a Qubit® 1.0 fluorometer and the Qubit® dsDNA HS assay (Life Technologies, Carlsbad). SOAPalign. SpecI (http://vmlux.embl.de/~kultima/MOCAT/) will be used to determine species composition and HUMAN (http://huttenhower.sph.harvard.edu/humann) used for the characterization of microbial pathways in the communities.
Serum metabolomics: Change is being assessed | Baseline, Week-8
  Metabolomics analysis provides a snapshot of an organism's current metabolite profile.blood serum samples will be prepared, including filtering and pH standardization and then all nuclear magnetic resonance (NMR) experiments performed on a Bruker Advance 600 spectrometer (Bruker Biospin, Milton, Canada). Processed spectra will be imported into Chenomx NMR Suite software (Edmonton, AB) for metabolite identification and quantification. metabolomics data will be integrated with the other biological variables assessed using O2PLS-DA
Health related quality of life: Change is being assessed | Baseline, Week-8
  Health-related quality of life will be measured using the 12-item short form-12. It comprises of two components physical health and mental Health. Scores range from 0 to 100, where a zero score indicates the lowest level of health and 100 indicates the highest level of health.
Dietary intake: Change is being assessed | Baseline, Week-8
  Dietary intake and supplement use will be assessed using two non-consecutive 24-hour food recalls using the ASA-24 Canadian version, and the Canadian Diet History II food frequency questionnaire (C-DHQ II). The non-consecutive 24-hour recalls will be used to calibrate the C-DHQ II. The ASA 24 is a freely available Web-based tool that enables automated self-administered 24-hour recalls. The C-DHQ II measures past month intake, includes portion sizes, and will be used to capture past month food intake
Physical Activity Monitoring: Change is being assessed | Baseline, Week-8
  Participants will be given a small device called 'Active Pal' at the baseline visit to monitor their physical activity for 7 days. They will be taught on wearing the device on their thigh for 7 days and return the device. Data will be extracted from the device and analyzed by the research team.
Cytokines Measurements: Change is being assessed | Baseline, Week-8
  IL-6, IL-10, NF-KB, TNF (tumor necrosis factor) alpha will be used to track inflammatory markers in the blood at baseline and week 8. Participants will be taken to get their blood taken during their baseline and 8 week appointments at the (Heritage Medical Research Clinic ) facility on the University of Calgary campus by the research coordinator.
Patient Survey Change is being assessed. | Baseline, Week-8
  Attitudes, social support, facilitators and barriers, and intention for changing dietary patterns using PDT will be measured using a Theory of Planned Behaviour survey.The Patient Assessment of Chronic Illness Care and 5A's survey (PACIC-5A)37,38 is a 26-item measure assessing chronic disease care from the patient perspective. It evaluates whether care was patient-centred, used appropriate behaviour counselling techniques, and connected patients to additional resources.

CONTACTS AND LOCATIONS:
Locations (1):
- TRW building, Foothills, University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Strauss JC, Haskey N, Ramay HR, Ghosh TS, Taylor LM, Yousuf M, Ohland C, McCoy KD, Ingram RJM, Ghosh S, Panaccione R, Raman M. Weighted Gene Co-Expression Network Analysis Identifies a Functional Guild and Metabolite Cluster Mediating the Relationship between Mucosal Inflammation and Adherence to the Mediterranean Diet in Ulcerative Colitis. Int J Mol Sci. 2023 Apr 15;24(8):7323. doi: 10.3390/ijms24087323. PMID 37108484